CLINICAL TRIAL: NCT04699903
Title: Clinical Evaluation of a Point-of-Care (POC), SARS-CoV-2 IgG Antibody Test in Fingerstick Whole Blood
Brief Title: Clinical Evaluation of a Point-of-Care (POC), SARS-CoV-2 (COVID-19) IgG Antibody Test in Fingerstick Whole Blood
Status: Completed | Type: Observational
Sponsor: Lumos Diagnostics (Industry)
Collaborators: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-1106
Record Dates: First submitted 2020-12-29; First posted 2021-01-07 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: SARS-Cov-2, Covid19
Keywords: IgG; Point of care testing; EUA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fingerstick whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Positive SARS-Cov-2 cohort: Positive diagnosis of COVID-19 confirmed by a positive EUA SARS-CoV-2 PCR will be stratified in three subgroups 0 - 7 days since onset of symptoms 8 - 14 days since onset of symptoms 15 -90 days since onset of symptoms
  Interventions: Diagnostic Test: POC SARS-Cov-2 IgG Antibody test
- Negative SARS-Cov-2 cohort: Negative diagnosis of COVID-19 confirmed by a negative, EUA SARS-CoV-2 PCR test within 0-7 days of PCR sample collection will be included in the negative cohort.
  Interventions: Diagnostic Test: POC SARS-Cov-2 IgG Antibody test

INTERVENTIONS:
Diagnostic Test: POC SARS-Cov-2 IgG Antibody test — All patients will undergo a Point of care (POC) SARS-Cov-2 IgG Antibody test in fingerstick whole blood

SUMMARY:
Prospective, multi-center, observational, blinded clinical trial to compare a new point of care (POC) SARS-CoV-2 IgG antibody test to a reference SARS-CoV-2 PCR test using fingerstick whole blood.

DETAILED DESCRIPTION:
Patients with PCR testing in outpatient setting will be screened and asked to participate in the study.

Subjects with a positive diagnosis of COVID-19 confirmed by a positive, EUA SARS-CoV-2 PCR test will be stratified by the number of days since first symptom onset (i.e. 0-7, 8-14, or >15 days) in the positive cohort Subjects with a negative diagnosis of COVID-19 confirmed by a negative, EUA SARS-CoV-2 PCR test within 0-7 days of PCR sample collection will be included in the negative cohort.

Treating clinicians, clinical research coordinators and study subjects will be blinded to the POC test results.

Quality assurance will be assured with site monitoring to check accuracy and completeness of data entered.

ELIGIBILITY:
Positive Cohort

Inclusion Criteria:

* Patients with high-sensitive EUA PCR results (positive result)
* Previous diagnostic of SARS-Cov-2
* Signed informed consent

Exclusion Criteria:

* Missing PCR results
* Results from a non-high-sensitive PCR test

Negative Cohort

Inclusion Criteria:

* Patients with high-sensitive EUA PCR results (negative result)
* Signed informed consent

Exclusion Criteria:

* Missing PCR results
* Results from a non-high-sensitive PCR test
* Previous diagnostic of SARS-Cov-2
* History of a positive SARS-CoV-2 antibody test (IgG, IgM or Total Antibody)
* Negative SARS-Cov-2 PCR result that occurred > 7 days from study visit

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the outpatient setting with EUA PCR test results who meet inclusion and exclusion criteria are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
PPA (positive percent agreement) and NPA (negative percent agreement) of POC compared to SARS-CoV-2 reference PCR | 0-7 days
  Determine PPA and NPA of point of care (POC) SARS-CoV-2 IgG antibody test compared to SARS-CoV-2 PCR with EUA (FDA emergency use authorization)
PPA (positive percent agreement) of POC compared to SARS-CoV-2 reference PCR | 8-14 days
  Determine PPA of point of care (POC) SARS-CoV-2 IgG antibody test compared to SARS-CoV-2 PCR with EUA (FDA emergency use authorization)
PPA (positive percent agreement) of POC compared to SARS-CoV-2 reference PCR | 15 - 90 days
  Determine PPA of point of care (POC) SARS-CoV-2 IgG antibody test compared to SARS-CoV-2 PCR with EUA (FDA emergency use authorization)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Benchmark - SoCal, Colton, California
  - Comprehensive Clinical Research, West Palm Beach, Florida
  - Great Lakes Clinical Trials (GLCT), Chicago, Illinois